CLINICAL TRIAL: NCT03068377
Title: The Effects of LycoRed Phytonutrient and Vitamin Supplement (a.k.a. LYC-001e) on Ocular Blood Flow
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LycoRed Ltd. (Industry)
Collaborators: Indiana University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: LYC-001e
Record Dates: First submitted 2017-02-26; First posted 2017-03-01 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Ocular Blood Flow
Keywords: lycopene; eye; vessel function

STUDY DESIGN:
Intervention Model Description: Single-phase, randomized, parallel, double blind , comparative study of LYC-001e versus placebo on ocular blood vessels in healthy individuals
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: randomized double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Soft gel capsules without test material
  Interventions: Dietary Supplement: Placebo
- Experimental (Experimental): Soft gel capsules containing a mixture of tomato extract, lutein, zeaxanthin as well as other phytonutrients and vitamins
  Interventions: Dietary Supplement: Experimental

INTERVENTIONS:
Dietary Supplement: Experimental — Soft gel capsules containing a mixture of tomato extract, lutein, zeaxanthin as well as other phytonutrients and vitamins
  Arms: Experimental
Dietary Supplement: Placebo — soft gel capsules without test material
  Arms: Placebo

SUMMARY:
Objectives:To determine LYC-001e's influences on ocular blood flow Ocular blood flow has been implicated as a parameter relevant to eye health and involved in the disease process of several ophthalmic pathologies including AMD, glaucoma, and diabetes We hypothesis that LYC-001e will increase measures of ocular blood flow in healthy individuals

Methods: This is a single-phase, randomized, parallel, double blind , comparative study of LYC-001e versus placebo on ocular blood vessels in healthy individuals.

DETAILED DESCRIPTION:
Age-Related Eye Disease (ARED) is a group of conditions that are associated with an increased risk of manifesting later in life, and include: Age-related Macular Degeneration (AMD), cataract, diabetic retinopathy, glaucoma, dry eye, and low vision. AMD and cataract are the leading causes of visual impairment in the United States. According to the National Eye Institute, approximately 1.7 million Americans suffer from some form of AMD, and over 1.5 million cataract surgeries are performed annually.

Although there are established risk factors, such as smoking and diabetes, cataracts are generally considered a consequence of ageing. The National Eye Institute estimates more than half of Americans will have cataracts or have had cataract surgery by the time they reach 80 years old. Additionally, AMD is the leading cause of central vision loss in developed countries and affects 13.4% of all adults aged 60 years and older.

It is estimated that the number of patients with AMD in the U.S. will double in 2050, based on 2010 demographics.

The severity and irreversibility of ocular pathology have created interest in researching ways to either prevent or slow their progression. Nutritional methods have been demonstrated to improve microvascular function in hypertensive patients, however diet modifications are infrequently well established and maintained in the American population.

Over the last 15 years, researchers focused on the role of the AREDS vitamin formulation on age related eye disease, specifically as it pertains to the development and progression of AMD and cataracts. While the benefit of AREDS supplementation has proven beneficial for AMD, its role in the prevention of cataract and/or glaucoma development has not been confirmed. However, with evidence suggesting that some combination supplements do provide potential risk reduction, it is our belief that further studies are needed to elucidate the role of combination nutriceuticals for the prevention of cataracts.

Lycored Nutrient Complex for eyes (LNC for eyes) a.k.a. (LYC-001e) is a commercially available multivitamin formula nutraceutical product that also contains a standardized tomato extract. Research by Armoza, et al. has shown multiple benefits of tomato extract as it pertains to limiting inflammatory processes of the vascular endothelium. Along with the previously mentioned benefits of nutraceuticals, diminished endothelial damage may result in increased ocular blood flow and alter the progression of Age Related Eye Diseases.

This is an important research consideration as ocular blood flow has been implicated in the disease process of several ophthalmic pathologies including AMD, glaucoma, and diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females of 18 years of age or older and free of any eye disease (other than myopia)
* Willing to sign an informed consent statement and able to comply with the requirements of the examination

Exclusion Criteria:

* Women who are pregnant or lactating or who plan to become pregnant (self reporting) within the duration of the study or within one month after study completion.

  * Receiving medications or dietary supplements known to have any interaction with the study supplements.
  * Smoker during last ten years (self reporting)
  * Concurrent use of any of the components of the study supplement
  * Individuals with narrow anterior chamber angles

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-03-20 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Retinal microcirculation via Heidelberg Retinal Flowmeter | 3 weeks
  Measures retinal capillary blood flow

SECONDARY OUTCOMES:
Ocular perfusion pressure | 3 weeks
  intraocular pressure and blood pressure
Retinal photographic oximetry | 3 weeks
  Measures oxygen content in retinal arteries and veins

CONTACTS AND LOCATIONS:
Overall Officials: Alon Harris, MS, PhD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Glaucoma Research and Diagnostic Center Eugene and Marilyn Glick Eye Institute Indiana University School of Medicine, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No